CLINICAL TRIAL: NCT02007083
Title: Comparison of Different Surgical Treatments for Lumbar Spinal Stenosis. A Randomized Controlled Trial Comparing the Clinical and Radiological Results Using "Spinous Process Osteotomy", "Bilateral Laminotomy" and "Unilateral Laminotomy With Crossover"
Brief Title: The NORDSTEN Studies/ The Spinal Stenosis Study
Acronym: NORDSTEN/SST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Møre og Romsdal Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011/2034; 2011/2034
Record Dates: First submitted 2013-11-22; First posted 2013-12-10 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Lumbar Spinal stenosis; Surgical treatment of LSS.
MeSH Terms: conditions — Spinal Stenosis | interventions — Crossing Over, Genetic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bilateral laminotomy (BL) (Active Comparator): The multifidus muscles is detached from the spinous process bilaterally.The decompression of the spinal canal is performed by first doing a flavectomy. Thereby performing a laminotomy (about 1/3) of the the lower part of the superior lamina, and a laminotomy of the upper part (about 1/4) of the inferior lamina. This is performed bilaterally.
  Interventions: Procedure: Bilateral laminotomy (BL)
- Unilateral laminotomy with crossover (UL) (Active Comparator): The multifidus muscles is detached from the spinous process unilaterally. The laminotomy is first performed ipsilaterally. The decompression of the spinal canal is performed by first doing a flavectomy. Then, performing a laminotomy (about 1/3) of the the lower part of the superior lamina, and a laminotomy of the upper part (about 1/4) of the inferior lamina. Dura is then retracted, and the decompression is performed contralaterally.
  Interventions: Procedure: Unilateral laminotomy with crossover (UL)
- Spinous process osteotomy (SPO) (Active Comparator): The multifidus muscles is detached from the spinous process unilaterally. An osteotomy of the superior spinous process is performed at the basis, in the actual level. The spinous process with intact interspinal and supraspinal ligaments is then retracted to the contralateral side. The decompression is first performed in the midline. Then one goes laterally on both sides too perform the decompression. About 1/3 of the lower part of the superior lamina is removed, and about 1/4 of the upper part of the inferior lamina is removed.
  Interventions: Procedure: Spinous Process Osteotomy (SPO)

INTERVENTIONS:
Procedure: Bilateral laminotomy (BL)
  Other Names: Fenestration procedures.; Multiple laminotomies.
  Arms: Bilateral laminotomy (BL)
Procedure: Unilateral laminotomy with crossover (UL)
  Other Names: microdecompression.
  Arms: Unilateral laminotomy with crossover (UL)
Procedure: Spinous Process Osteotomy (SPO)
  Other Names: Laminarthrectomi.; Micro Spinous Process Osteotomy
  Arms: Spinous process osteotomy (SPO)

SUMMARY:
Lumbar Spinal Stenosis (LSS) is a clinical entity were narrowing of the spinal canal gives a compression of the the neural and vascular structures in the spinal canal. This often gives neurogenic claudication and sometimes severe Low Back Pain (LBP). Surgery for LSS is today the most often performed procedure in the adult lumbar spine. Beneficial effect of surgical treatment is well documented by several clinical trials, and a Cochrane review article from 2005 concludes that surgical treatment is superior to non-surgical treatment. The surgical solution is to decompress the stenotic part of the lumbar spine. There is no consensus in the literature of which surgical method that gives best long term clinical results. The investigators are therefore planning a Randomized Controlled Trial, where they will compare clinical and radiological results of three different surgical methods for LSS. The main outcome of this study is to answer which surgical method that gives the best long term clinical results. And, secondary outcome is to find out how much increase of the Dural Sac Cross Sectional Area is needed to give a long time relief of the patients' symptoms.

ELIGIBILITY:
Inclusion Criteria:

* have clinical symptoms of spinal stenosis as neurogenic claudication or radiating pain into the bilaterally to the lower limbs, not responding to at least 3 months of conservative treatment.
* Radiological findings corresponding to the clinical symptoms of LSS. Central -stenosis, or lateral recess-stenosis.
* be able to give informed consent and to answer the questionnaires.
* over 18 years of age-have -not responding to at least 3 months of non-surgical treatment.
* be able to understand Norwegian language, spoken and in writing

Exclusion Criteria:

* have a degenerative lumbar spondylolisthesis, with a slip ≥ 3 mm verified on standing plain x-rays in lateral view.
* are not willing to give written consent.
* have former surgery in the level of stenosis.
* fracture, or former fusion of the thoracolumbal region.
* cauda equina syndrome (bowel or bladder dysfunction) or fixed complete motor deficit.
* are ASA- classified 4 or 5.
* are older than 80 years
* have a lumbosacral scoliosis more than 20 degrees verified on AP-view
* have distinct symptoms in one or both of their legs due to other diseases, e.g. polyneuropaty, vascular claudication or osteoarthtris.
* LSS in 4 or more levels.
* not able to comply fully with the protocol, including treatment, follow-up or study procedures (psychosocially, mentally and physical).
* the patient is participating in another clinical trial that may interfere with this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Estimated)
Dates: Start 2013-11 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index | 2, 5 and 10 years after surgery
  The investigators will monitor the ODI-index before and after surgery, and calculate the change of ODI after surgery compared to baseline.
  The primary outcome is a measurement of the change of ODI (version 2.0) from baseline in the three different surgical groups. This will be done by calculating the mean ODI improvement in each group. The investigators will also compare the proportion of "success patients" between the SPO group, the BL group and the UL group, 24 months after the operation. The investigators will dichotomize the patients, in a "succesful outcome group" and in a "non- succesful outcome group". The threshold value for being categorized as a "succesful outcome" will be computed in a planned study based on data from The Norwegian Registry for Spine Surgery (NORSpine).
  The investigators also plan to asses short time results after 2 years, intermediate results after 5 years, and long time results after 10 years.

SECONDARY OUTCOMES:
Zurich claudification Scale, Numeric Rating Scale for leg pain, Numeric Rating Scale for back pain, EQ-5D, and self evaluated effect of surgery. | 2, 5 and 10 years after surgery
  All of the above mentioned questionaires are validated and reliable questionaires to asses the effect of surgical treatment. The effect of the surgical treatment is calculated by the improvement of the different scores, and thereby is an objective way to asses the effect of the surgical treatment.
  The investigators plan to asses short time results after 2 years, intermediate results after 5 years, and long time results after 10 years.

OTHER OUTCOMES:
Dural Sac Cross sectional Area (DSCSA) | 3 months after surgery
  The investigators are planning to investigate the DSCSA before and after surgery. Thereby we can monitor which surgical procedure that increases the DSCSA the most. The investigators will also investigate wether a large increase of the DSCSA is needed to maintain good long-time clinical results.

CONTACTS AND LOCATIONS:
Overall Officials: Kari Indrekvam Indrekvam, MD, Dr Med, Study Director — The Coastal Hospital of Hagevik, Orthopeadic Clinic, Haukeland University City
Locations (1):
- Haukeland University Hospital, Bergen, Hagevik, Norway

REFERENCES:
- [Derived] Indrekvam K, Myklebust TA, Austevoll IM, Hermansen E, Banitalebi H, Banerud IF, Weber C, Brisby H, Brox JI, Hellum C, Storheim K. Responsiveness of the Oswestry Disability Index and Zurich Claudication Questionnaire in patients with lumbar spinal stenosis: evaluation of surgically treated patients from the NORDSTEN study. Eur Spine J. 2024 Nov;33(11):4270-4280. doi: 10.1007/s00586-024-08440-1. Epub 2024 Aug 13. PMID 39134699
- [Derived] Aaen J, Banitalebi H, Austevoll IM, Hellum C, Storheim K, Myklebust TA, Anvar M, Weber C, Solberg T, Grundnes O, Brisby H, Indrekvam K, Hermansen E. Is the presence of foraminal stenosis associated with outcome in lumbar spinal stenosis patients treated with posterior microsurgical decompression. Acta Neurochir (Wien). 2023 Aug;165(8):2121-2129. doi: 10.1007/s00701-023-05693-5. Epub 2023 Jul 5. PMID 37407851
- [Derived] Indrekvam K, Banerud IF, Hermansen E, Austevoll IM, Rekeland F, Guddal MH, Solberg TK, Brox JI, Hellum C, Storheim K. The Norwegian degenerative spondylolisthesis and spinal stenosis (NORDSTEN) study: study overview, organization structure and study population. Eur Spine J. 2023 Dec;32(12):4162-4173. doi: 10.1007/s00586-023-07827-w. Epub 2023 Jul 3. PMID 37395780
- [Derived] Hermansen E, Austevoll IM, Hellum C, Storheim K, Myklebust TA, Aaen J, Banitalebi H, Anvar M, Rekeland F, Brox JI, Franssen E, Weber C, Solberg TK, Furunes H, Grundnes O, Brisby H, Indrekvam K. Comparison of 3 Different Minimally Invasive Surgical Techniques for Lumbar Spinal Stenosis: A Randomized Clinical Trial. JAMA Netw Open. 2022 Mar 1;5(3):e224291. doi: 10.1001/jamanetworkopen.2022.4291. PMID 35344046
- [Derived] Banitalebi H, Espeland A, Anvar M, Hermansen E, Hellum C, Brox JI, Myklebust TA, Indrekvam K, Brisby H, Weber C, Aaen J, Austevoll IM, Grundnes O, Negard A. Reliability of preoperative MRI findings in patients with lumbar spinal stenosis. BMC Musculoskelet Disord. 2022 Jan 15;23(1):51. doi: 10.1186/s12891-021-04949-4. PMID 35033042
- [Derived] Aaen J, Austevoll IM, Hellum C, Storheim K, Myklebust TA, Banitalebi H, Anvar M, Brox JI, Weber C, Solberg T, Grundnes O, Brisby H, Indrekvam K, Hermansen E. Clinical and MRI findings in lumbar spinal stenosis: baseline data from the NORDSTEN study. Eur Spine J. 2022 Jun;31(6):1391-1398. doi: 10.1007/s00586-021-07051-4. Epub 2021 Nov 19. PMID 34797405
- [Derived] Hermansen E, Austevoll IM, Hellum C, Storheim K, Myklebust TA, Aaen J, Banitalebi H, Anvar M, Rekeland F, Brox JI, Franssen E, Weber C, Solberg T, Haug KJ, Grundnes O, Brisby H, Indrekvam K. Comparable increases in dural sac area after three different posterior decompression techniques for lumbar spinal stenosis: radiological results from a randomized controlled trial in the NORDSTEN study. Eur Spine J. 2020 Sep;29(9):2254-2261. doi: 10.1007/s00586-020-06499-0. Epub 2020 Jun 18. PMID 32556585
- [Derived] Hermansen E, Austevoll IM, Romild UK, Rekeland F, Solberg T, Storheim K, Grundnes O, Aaen J, Brox JI, Hellum C, Indrekvam K. Study-protocol for a randomized controlled trial comparing clinical and radiological results after three different posterior decompression techniques for lumbar spinal stenosis: the Spinal Stenosis Trial (SST) (part of the NORDSTEN Study). BMC Musculoskelet Disord. 2017 Mar 21;18(1):121. doi: 10.1186/s12891-017-1491-7. PMID 28327114